CLINICAL TRIAL: NCT01870219
Title: The Effects of Sevoflurane or Ketamine on QTc Interval During Electroconvulsive Therapy
Brief Title: Effects of Sevoflurane and Ketamine on QT in Electroconvulsive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Feray Erdil, MD, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Turgut Ozal Medical Center
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Major Depression; Electroconvulsive Therapy
Keywords: sevoflurane; ketamine; QT interval
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sevoflurane; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group S (Active Comparator): In group S, sevoflurane was initiated at %8 sevoflurane for anesthesia induction and maintained at 2% to %4 until the electrical stimulus was delivered, at which time it was turned off.
  Interventions: Drug: Sevoflurane
- Group K (Active Comparator): In group K, ketamine was given to 1mg/kg ıv bolus.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Sevoflurane — sevoflurane was initiated at %8 sevoflurane for anesthesia induction and maintained at 2% to %4 until the electrical stimulus was delivered
  Other Names: Volatile agent
  Arms: Group S
Drug: Ketamine — ketamine was given to 1mg/kg ıv bolus
  Other Names: Intravenous anesthetic agent
  Arms: Group K

SUMMARY:
The aim of this study was to evaluate the effect of sevoflurane or ketamine on the QTc and Tp-e interval during in patients with major depression.

DETAILED DESCRIPTION:
Patients enrolled in the study are randomly allocated by computer-generated random numbers to receive either sevoflurane or ketamine for their initial ECT session. They subsequently receive an alternative study drug in their next session, continuing to alternate between drugs at each session until the sixth session. In group S, sevoflurane are initiated at %8 sevoflurane for anesthesia induction and maintained at 2% to %4 until the electrical stimulus is delivered, In group K, ketamine are given to 1mg/kg ıv bolus.

Electrical stimulus is delivered via bilateral frontotemporal electrodes.The mean arterial pressure (MAP), HR, and ECG are recorded before anesthetic induction (T1), after anesthetic induction (T2) and at 0, 1, 3, 10 min after the seizure ended (T3, T4, T5 and T6, respectively).The QT interval and Tp-e interval are measured by one author, who was unaware of group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Unpremedicated
* American Society of Anesthesiologists (ASA) I-II the patients
* Major depressions patients scheduled for ECT sessions

Exclusion Criteria:

* pregnant
* with permanent pacemakers,
* diabetes mellitus,
* atrial fibrillation,
* electrolyte imbalance,
* patients taking antiarrhythmics and β-blockers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Evaluation Of QT interval | 10 minutes
  ECG were recorded before anesthetic induction (T1), after anesthetic induction (T2) and at 0, 1, 3, 10 min after the seizure ended (T3, T4, T5 and T6, respectively)during ECT anesthesia with sevoflurane and ketamine.The QT interval was measured by one author, who was unaware of group allocation.

SECONDARY OUTCOMES:
Evaluation of Tp-e interval | 10 minutes
  ECG were recorded before anesthetic induction (T1), after anesthetic induction (T2) and at 0, 1, 3, 10 min after the seizure ended (T3, T4, T5 and T6, respectively)during ECT anesthesia with sevoflurane and ketamine.The Tp-e interval was measured by one author, who was unaware of group allocation.
Seizure durations | 120 seconds
  The duration of the EEG seizure was recorded from the EEG trace, and the peak heart rate (HR) during the convulsion was recorded from the ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Feray Erdil, MD, Principal Investigator — Associated Prof Dr
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Erdil F, Demirbilek S, Begec Z, Ozturk E, Ersoy MO. Effects of propofol or etomidate on QT interval during electroconvulsive therapy. J ECT. 2009 Sep;25(3):174-7. doi: 10.1097/YCT.0b013e3181903fa5. PMID 19225403